CLINICAL TRIAL: NCT02595801
Title: Surgery in Early Life and Child Development at School-entry: A Population-based Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: McMaster University (Other); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, James O'Leary, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000046454
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Surgery in Early Childhood
MeSH Terms: interventions — Surgical Procedures, Operative; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Exposed: Exposure to surgery prior to completion of Early Development Instrument
  Interventions: Other: Surgery in early childhood
- Reference: No exposure to surgery prior to completion of Early Development Instrument

INTERVENTIONS:
Other: Surgery in early childhood — Surgical interventions in early childhood (prior to completion of Early Development Instrument)
  Other Names: Surgery/Anesthesia in early childhood
  Groups: Exposed

SUMMARY:
The central hypothesis is that surgery and anesthesia exposure in children with immature structural and functional brain development has long-term adverse effects on child development at school-entry compared with children not exposed to anesthesia.

The secondary hypothesis is that frequency of surgery and anesthesia exposure in children with immature structural and functional brain development has a dose-dependent association with worsened child development outcomes at school-entry.

The overall objective is to investigate the association between surgery/anesthesia exposure(s) in children in Ontario and major child development outcomes (physical health and well being, social competence, emotional maturity, and language and cognitive development) at school entry as measured by the Early Development Instrument.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Early Development Instrument in Ontario

Exclusion Criteria:

* Children with physical or developmental disabilities identified in the Early Development Instrument
* Not born in Canada
* Having undergone fetal interventions, radiation or brachytherapy, local pharmacotherapy, systemic cancer chemotherapeutic procedures, therapeutic interventions of the cardiovascular system
* Patients of a cardiology or cardiovascular service

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children attending public or Catholic school in Ontario who have completed the Early Development Instrument
Sampling Method: Non-Probability Sample
Enrollment: 188628 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Early developmental vulnerability | Assessed between five and six years of age
  Any major domain of the Early Development Instrument in the lowest 10th percentile

SECONDARY OUTCOMES:
Performance in specific Early Development Instrument domains | Assessed between five and six years of age
  Vulnerability (percentage in lowest 10th centile); mean score
Multiple challenge index | Assessed between five and six years of age
  Vulnerability (percentage in lowest 10th centile) in ≥9 sub-domains of the Early Development Instrument

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada